CLINICAL TRIAL: NCT01367275
Title: Phase II Study of Second-line Irinotecan Plus Brivanib, a Dual Tyrosine Inhibitor of VEGFR and FGFR, in Metastatic Colorectal Cancer Patients Enriched for Elevated Levels of Plasma FGF Following Progression on Bevacizumab-based Treatment
Brief Title: Irinotecan Plus Brivanib in Metastatic Colorectal Cancer (CRC) Enriched for Elevated Levels of Plasma FGF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor closed study
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0378
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma
Keywords: colon; Colorectum; Colorectal Cancer; Plasma FGF; Colorectal adenocarcinoma; Bevacizumab; Brivanib; BMS-582664; Irinotecan; CPT-11; Camptosar; Fibroblast Growth Factor; bFGF; tyrosine kinase receptors; vascular endothelial growth factor receptors; VEGFR; fibroblast growth factor receptors; FGFR
MeSH Terms: conditions — Colorectal Neoplasms; Acrocephalosyndactylia | interventions — brivanib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivanib + Irinotecan (Experimental): Brivanib 800 mg orally daily Days 1-14, and Irinotecan intravenously 180 mg/m^2 on Day 1.
  Interventions: Drug: Brivanib; Drug: Irinotecan

INTERVENTIONS:
Drug: Brivanib — 800 mg (4 x 200 mg tablets) self-administered orally at approximate same time each day on a continuous daily schedule Days 1-14 of 14 day cycle.
  Other Names: BMS-582664
Drug: Irinotecan — 180 mg/m^2 by vein on Day 1 of a 14 day cycle.
  Other Names: CPT-11; Camptosar

SUMMARY:
The goal of this clinical research study is to learn if adding brivanib to irinotecan can help control the disease in patients with colorectal cancer that has spread. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Brivanib is designed to keep cancer cells from receiving the blood supply they need. This may slow down the growth of cancer cells.

Irinotecan is designed to interfere with the DNA (genetic material) of cancer cells. This may slow down the growth and spread of cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take brivanib by mouth 1 time every day. The study drug should be taken at the same time each day with a glass (about 8 ounces) of water. You can take it with or without food.

You will be given irinotecan by vein over about 1½ hours on Day 1 of each 14-day cycle. You may be given other drugs to help prevent side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

If you have a side effect, you should tell your doctor or study nurse right away. Your study doctor may prescribe drugs for your side effects, delay future treatments, lower the dose of the study drugs, or stop your treatment with the study drugs.

Study Visits:

On Day 7 of Cycle 1:

* Your vital signs will be measured.
* Blood (about 2 tablespoons) will be drawn for routine tests and to check your thyroid function. If the doctor thinks it is needed, part of the blood may be used to check your blood's ability to clot.

Before all cycles, starting with Cycle 2:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 1-2 tablespoons) will be collected for routine tests. If the doctor thinks it is needed, part of the blood may be used to check your blood's ability to clot if needed.
* You will be asked about any drugs you may have taken and side effects you may have had.
* Before Cycles 2 and 3 only, blood (about 1 tablespoon) will be drawn to check your thyroid function.

Every 8 weeks:

* You will have a CT scan or MRI scan to check the status of the disease.
* Blood (about 2-3 tablespoons) will be drawn for thyroid, CEA, and cytokine testing.
* Urine will be collected for routine tests.

Every 12 weeks (Weeks 12, 24, 36, and so on), you will have an ECHO to check your heart function.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

End-of-Treatment Visit:

Within 2 weeks after you stop taking the study drugs, the following tests and procedures will be performed if not done in the last 14 days:

* You will be asked about any side effects you may have had and any drugs you may be taking.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will have a CT scan or MRI scan to check the status of the disease.
* Blood (about 1-2 tablespoons) and urine will be collected for routine tests.
* Blood (about 2-3 tablespoons) will be drawn for thyroid, CEA, and cytokine testing.

Long-Term Follow-Up:

After you stop taking the study drugs, you will be called every 3 months. You will be asked questions about your health. These calls should last about 15 minutes each time.

This is an investigational study. Brivanib is not FDA approved or commercially available. It is currently being used for research purposes only. Irinotecan is FDA approved and commercially available for the treatment of colorectal cancer. The combination of brivanib and irinotecan is considered investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent.
2. Patient must have progressed on front-line chemotherapy treatment containing bevacizumab for histologically confirmed colorectal adenocarcinoma that is unresectable or metastatic. Progression is defined as either radiographic or clinical progression.
3. Patient must have measurable lesions as defined by RECIST version 1.1 criteria.
4. ECOG performance status 0-2.
5. Known bFGF level performed by a CLIA-certified laboratory performed during or within 12 weeks of last bevacizumab treatment
6. Enrollment in the "Assessment of Targeted Therapies Against Colorectal Cancer" (ATTACC) protocol 2009-0091.
7. LVEF > 50% measured by 2-D echocardiogram
8. Bone marrow function defined as the following: An absolute neutrophil count (ANC) =/>1,500/mcl; Platelets =/>100,000/mcl; Hemoglobin =/> 8.5 g/dl.
9. Renal function defined as the following: Serum creatinine less than or equal to 1.5 x institutional upper limit normal (ULN).
10. Hepatic function defined as the following: Serum total bilirubin < 1.5 x ULN; AST (SGOT), ALT (SGPT) and alkaline phosphatase =/< 2.5 x ULN; Serum albumin =/> 2.5 g/dl; If liver involvement, AST, ALT, and alkaline phosphatase =/< 5.0 x ULN.
11. International normalized ratio (INR) =/< 2.3 or Prothrombin Time (PT) =/< 6 seconds above control unless patient is currently receiving warfarin therapy for the treatment or prevention of venous thrombosis.
12. Men and women, age =/> 18 years.
13. A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study [and for up to 12 weeks after the last dose of study drug] to minimize the risk of pregnancy. If the partner is pregnant or breastfeeding, the subject must use a condom.
14. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy. WOCBP must have a negative serum or urine pregnancy test within 72 hours before the start of the investigational product.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Patients with brain metastases.
3. Patients with resectable colorectal cancer or non-adenocarcinoma cancer of the colon or rectum.
4. Patients who have had prior therapy with brivanib, anti-PDGFR (platelet-derived growth factor receptor) or anti-FGFR (fibroblast growth factor receptor) therapy.
5. Recent (within 4 weeks of the first study drug administration), or planned participation in another experimental therapeutic drug study.
6. Recent (within 4 weeks of the first study drug administration) infusion of bevacizumab therapy.
7. Prior irinotecan chemotherapy.
8. Prior full field radiotherapy =/<4 weeks or limited field radiotherapy =/<2 weeks prior to first study drug administration.
9. Recent use (within 4 weeks of first study drug administration) of St. John's Wort.
10. Patients with a history of thrombotic or embolic events within the last six months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism.
11. Patients with gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE (version 4.0) Grade 4 within 30 days prior to first study drug administration
12. Patients with uncontrolled or significant cardiovascular disease including: i) Active coronary artery disease, unstable or newly diagnosed angina or myocardial infarction < 12 months prior to first study drug administration. ii) Class III-IV New York Heart Association (NYHA) congestive heart failure. iii) Uncontrolled hypertension (Systolic blood pressure [BP] > 150 mmHg and diastolic BP > 90 mmHg for 24 hours) despite optimal medical management. Blood pressure must be below 140/90 mmHg at screening. Subjects with a history of hypertension who are receiving treatment with calcium channel blockers that are CYP3A4 substrates should be changed to an alternative antihypertensive medication prior to first study drug administration. iv) Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin. v) QTc (Fridericia) prolongation >450 msec. vi) Subjects with valvular heart disease =/> CTCAE (Ver. 4.0) Gr 2. vii) Left ventricular ejection fraction (LVEF) < 50%.
13. Active infection, less than 7 days after completing systemic antibiotic therapy.
14. History of non-healing wounds or ulcers, or bone fractures within 3 months prior to first study drug administration.
15. Major surgical procedure, open biopsy, or significant traumatic injury less than 3 weeks or those who receive minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 1 week from first dose of first study drug administration.
16. Inability to swallow tablets or untreated malabsorption syndrome.
17. Pre-existing thyroid abnormality with thyroid function that can not be maintained in the normal range with medication.
18. History of human immunodeficiency virus (HIV).
19. Patients with centrally cavitating lung lesions.
20. Known bleeding diathesis.
21. Inability to comply with study and/or follow-up procedures.
22. Patients with known glomerular nephritis.
23. Patients with known polycythemia.
24. Patients with known Gilbert's syndrome.
25. Women with a positive pregnancy test.
26. Patients with hyponatremia (sodium < 130 mmol/L).
27. Baseline serum potassium < 3.5 mmol/L (potassium supplementation may be given to restore the serum potassium above this level prior to study entry).
28. Baseline serum calcium < 8.4 mg/dL (calcium supplementation may be given to restore the serum calcium above this level prior to study entry).
29. Baseline serum magnesium < 1.5 mg/dL (magnesium supplementation may be given to restore the serum magnesium above this level prior to study entry).
30. Known or suspected history of allergy to brivanib or any agents given in association with this study.
31. Prisoners or subjects who are involuntarily incarcerated. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 16, 2011 to September 7, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Early termination due to drug sponsor decision to no longer develop drug. One participant was enrolled but not eligible therefore not treated.
Groups:
- Brivanib + Irinotecan: Brivanib 800 mg orally daily Days 1-14, and Irinotecan intravenously 180 mg/m^2 on Day 1. One cycle is 14 days.
Period: Overall Study
Arm/Group | Brivanib + Irinotecan
Started | 8
Completed | 5
Not Completed | 3
Not completed — Ineligible | 1
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Population: Study was terminated early by sponsor with low accrual. Due to small number of participants, no statistical analysis was possible.
Arm/Group | Brivanib + Irinotecan
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 55 [43 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Median Progression-Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Enrollment (baseline) to disease progression or death, followed each 14 day treatment then every 2 months,up to 100 week
Measure: Count of Participants; unit: Participants
Arm/Group | Brivanib + Irinotecan
Number analyzed (Participants) | 8
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each 14 day treatment cycle and following two weeks after the last treatment, for up to 72 weeks.
Description: One participant enrolled of the eight (8) was not treated, therefore seven (7) participants are reported as the at risk population.
Arm/Group | Brivanib + Irinotecan
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivanib + Irinotecan (N=7)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivanib + Irinotecan (N=7)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Anal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (5)
Bloating (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (15)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Fever (General disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Mouth Sores, Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Fall, general soreness (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (5)
Colitis (Infections and infestations) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 6 (11)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2)
Pain (gluteal region) (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7)
Weight loss (Investigations) | 1 (8)
White blood cell decreased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
As a result of the drug sponsor closing study early, the accrual goal was not met and with the small number of participants enrolled no statistical analysis or conclusions was possible from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes